CLINICAL TRIAL: NCT07403253
Title: Comparative Effects of Fascial Distortion Model and Hamstring Stretching on Pain, Muscle Flexibility and Physical Function in Patients With Knee Osteoarthritis.
Brief Title: Comparative Effects of Fascial Distortion Model and Hamstring Stretching in Patients With Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/01106
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; hamstring tightness; hamstring stretching; fascial distortion model
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascial Distortion Model (Experimental)
  Interventions: Other: Fascial Distortion Model; Other: Standardize Physiotherapy Treatment
- Hamstring Stretching (Active Comparator)
  Interventions: Other: Hamstring Stretching; Other: Standardize Physiotherapy Treatment

INTERVENTIONS:
Other: Fascial Distortion Model — Put direct pressure on the fascia's taut band. The pressure should be just right, firm enough to activate the tissue without causing undue pain or discomfort. The pressure is usually extended across the bands length, or perpendicular to the direction of the band's fibers. Each stroke of the treatment might take between 10 to 30 seconds, depending on the severity of fascial distortion. A typical rule is to work through the band gently and consistently, without rushing, to allow the tissues time to respond. Treatment might be applied for 5 to 10 minutes, 2-3 times per week for 4 weeks
  Arms: Fascial Distortion Model
Other: Hamstring Stretching — With your legs relaxed and straight, lie on your back. Wrap a towel or strap under your foot arch, around your hamstring, or around your calf. Pull your leg gently in your direction until it stretches. It also entails stretching with the aid of an outside force, such as gravity or a partner. This position was held for 30 seconds, for 3 sets per sessions, 3 times in a week for 4 weeks
  Arms: Hamstring Stretching
Other: Standardize Physiotherapy Treatment — Hot pack for 10 minutes. TENS with frequency of 2Hz and pulse duration of 50-200 μs for 10 minutes and Knee strengthening exercise consists of (Isometric quadriceps strengthening exercise, straight leg raises, partial squatting exercise, knee extensor strength exercise) 10 repetition per set, 3 sets per sessions, 3 times in a week for 4 weeks.

SUMMARY:
The study was conducted to compare the effects of Fascial Distortion Model and Hamstring Stretching on pain, muscle flexibility and physical function in patients with Knee Osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Patient aged 40-60 years old of both genders.
  * X-ray showing unilateral degenerative changes in Knee joint.
  * Knee osteoarthritis stage 2 and stage 3 was included.
  * A score of 3 to 7 on the numeric pain rating scale (NPRS).
  * Patients with positive 90-90 hamstring flexibility test by using goniometer.

Exclusion Criteria:

* Recent fracture.
* The participants with any neurological disorder that impacts the lower extremity, Musculoskeletal knee deformity e.g. varus or valgus knee deformity, lower limb internal fixation etc .
* History of lower limb arthroplasty or knee surgery.
* Patients with body mass index (BMI) more than 35 were excluded.
* Previous history of malignancy or any infectious disease.
* Subjects having sciatica or low back pain were excluded from the study .

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC): | from enrollment to the end treatment of 4 weeks
  It is frequently used to assess osteoarthritis in the knee and hips. It is self- administered survey with three subscales and 24 items:
  * Pain (5 items): walking, climbing stairs, lying down or sitting, lying in bed and standing up straight.
  * Physical function (17 items): using stairs, getting up from sitting, standing, bending, walking, getting in and out of car, shopping, putting on or taking off socks, getting in and out of a bath, sitting, getting on and off the toilet, heavy domestic duties, and light domestic duties.
  * Stiffness (2 items): after first waking and later in the day. A possible score ranges of 0-20 for pain, 0-8 for stiffness and 0-68 for physical function is obtained by adding the score for each subscale. The overall WOMAC score ranges from 0-96, with 0 denoting the highest potential for health and 96 the worst. The function is worse, the higher the score.
Numeric Pain Rating Scale (NRRS) | from enrollment to the end of treatment at 4 weeks
  The NPRS was used to gauge the patient's degree of pain. On a 0-10 scale, where 0 represents no pain, 1-3 represents mild pain, 4-6 represents moderate pain, 7-10 represents severe pain, this tool is frequently used to gauge the intensity of pain. Patients rate how much pain they are currently experiencing as well as how much pain they had experienced in the past 24 hours. The patient's level of pain may be represented by average of the three evaluations or by any one rating. NPRS reliability is 0.96 and validity is 0.86.
90 -90 HAMSTRING FLEXIBILITY TEST | from enrollment to the end of treatment of 4 weeks
  The individual is in supine position with their arms folded across their chest their head back. If a spirit level is available, use it to passively flex the hi until the thigh is vertical. Throughout the test, keep the opposing leg fully extended while maintaining this thigh position. The leg being tested is actively straightened until the thigh starts to deviated from the vertical position, while the foot is kept relaxed. At this point, the thigh angle is noted. When the thigh is vertical, measure the minimum angle of knee flexion. Degrees are the unit of measurement. The angle would be reported as 0 if the leg could be fully straightened. Any amount of flexion, such as 10 to 20 degrees, will be noted as a positive number. Muscle tension is indicated by a value greater than 20 degrees. The knee is flexed the thigh is pushed 30 degrees past in the vertical position and the knee is straightened once more in situation where complete knee extension is accomplished without thigh movement.

SECONDARY OUTCOMES:
Knee Flexion ROM | from enrollment to the end of treatment at 4 weeks
  Changes in knee flexion ROM at baseline and 4th week of intervention was measured using goniometer.
Knee Extension ROM | From enrollment to the end of treatment at 4 weeks
  Changes in knee extension ROM at baseline and 4th week of intervention was measured using goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Rafia Mannan, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Abdul Ahaad hospital, Sialkot., Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahmoud, W.S., et al., Radiological and clinical outcomes of concurrent hamstring stretching with quadriceps strengthening in patients with knee osteoarthritis: A randomized clinical trial. Isokinetics and Exercise Science, 2023. 31(2): p. 137-147.